CLINICAL TRIAL: NCT01735422
Title: A Phase II, Single Center, Open, Randomized, Parallel Group, Dose Finding Study to Assess the Safety and Efficacy of Recombinant Human Luteinizing Hormone (r-hLH), Compared With Urinary Human Chorionic Gonadotrophin (u-hCG), in Inducing Ovulation in Infertile Women Undergoing Stimulation of Follicular Development With Recombinant Human Follicle Stimulating Hormone (Gonal F®).
Brief Title: A Study to Evaluate Safety and Efficacy of Recombinant Human Luteinizing Hormone (r-hLH) Compared With Urinary Human Chorionic Gonadotrophin (u-hCG) to Trigger Ovulation in Infertile Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21321
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Infertility
Keywords: Infertility; Ovulation induction; Recombinant human Luteinizing Hormone (r-hLH); Urinary human Chorionic Gonadotrophin (u-hCG); Recombinant human Follicle Stimulating Hormone (Gonal-f®)
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- r-hLH (825 International Units [IU]) (Experimental)
  Interventions: Drug: r-hFSH; Drug: r-hLH
- r-hLH (2750 IU) (Experimental)
  Interventions: Drug: r-hFSH; Drug: r-hLH
- r-hLH (5500 IU) (Experimental)
  Interventions: Drug: r-hFSH; Drug: r-hLH
- r-hLH (11000 IU) (Experimental)
  Interventions: Drug: r-hFSH; Drug: r-hLH
- r-hLH (22000 IU) (Experimental)
  Interventions: Drug: r-hFSH; Drug: r-hLH
- u-hCG (5000 IU) (Active Comparator)
  Interventions: Drug: r-hFSH; Drug: u-hCG

INTERVENTIONS:
Drug: r-hFSH — Daily r-hFSH treatment will be administered subcutaneously at a starting dose according to the site's standard practice from Day 3-5 of menstrual cycle up to follicular development or 28 days. Dose can be altered according to ovarian response (reduced to 75 IU/day; increased to 225 IU/day).
  Other Names: Gonal-f®
Drug: r-hLH — Ovulation triggering will be performed using a single injection of r-hLH injection subcutaneously at a dose of 825 or 2750 or 5500 or 11,000 or 22,000 IU as soon as follicles satisfy the criteria for follicular development, that is at least 1 follicle with diameter >= 18 mm, not more than 5 follicles with diameter >= 15 mm and with E2 levels less than 9000 picomoles per liter (pmol/L).
  Other Names: LHadi®
  Arms: r-hLH (11000 IU); r-hLH (22000 IU); r-hLH (2750 IU); r-hLH (5500 IU); r-hLH (825 International Units [IU])
Drug: u-hCG — Ovulation triggering will be performed using a single injection of 5000 IU of u-hCG as soon as follicles satisfy the criteria for follicular development, that is at least 1 follicle with diameter >= 18 mm, not more than 5 follicles with diameter >= 15 mm and with E2 levels less than 9000 picomoles per liter (pmol/L).
  Arms: u-hCG (5000 IU)

SUMMARY:
This is a single center, open-label, randomized, parallel group, dose finding study to evaluate safety and efficacy of recombinant human luteinizing hormone (r-hLH, LHadi®), compared with urinary human chorionic gonadotrophin (u-hCG, Profasi®), both given subcutaneously, in inducing ovulation in infertile women undergoing stimulation of follicular growth with recombinant human follicle stimulating hormone (r-hFSH, Gonal-F®).

ELIGIBILITY:
Inclusion Criteria:

* Infertile woman wishing to conceive and justifying ovarian stimulation treatment with gonadotrophins for in vivo conception
* Aged 20-40 years (inclusive)
* Male partner with acceptable semen analysis for intra-uterine insemination, according to center's standard practice
* Have the following hormone serum levels measured locally during early (Day 2-4) follicular phase (if menstruating) or at anytime (if not menstruating):

  * Follicle stimulating hormone (FSH) less than 12 international unit per liter (IU/L)
  * Prolactin (PRL) less than 800 milli international unit per liter (mIU/l)
  * Lutenizing hormone (LH), P4, Testosterone (T) and Dehydroepiandrosterone sulphate (DHEA-S) for documentation purposes
* At least one patent tube, as assessed with hysterosalpingography (HSG), ultrasound (U/S) or laparoscopy performed within 3 years prior to beginning r-hFSH treatment
* Uterine cavity without abnormalities which, in the Investigator's opinion, could impair embryo implantation or pregnancy evolution as assessed with HSG, hysteroscopy (HSC) or U/S performed within 3 years prior to beginning r-hFSH treatment
* Body mass index (BMI) greater than or equal to 18 and less than or equal to 35 kilogram per square meter (kg/m^2)
* Negative serum or urinary pregnancy test prior to beginning r-hFSH treatment
* Be willing and able to comply with the protocol for the duration of the study
* Have given written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care

Exclusion Criteria:

* Any contraindication to being pregnant and/or carrying a pregnancy to term
* Clinically significant systemic disease (screening for Human Immunodeficiency Virus (HIV) and Hepatitis B and C surface antigens had to be performed to confirm eligibility, unless data obtained within one year prior to beginning r-hFSH treatment was available)
* Any medical condition which in the judgment of the Investigator's and sponsor may have interfered with the absorption, distribution, metabolism or excretion of the study drug
* Persistent ovarian cyst with a mean diameter larger than 20 mm or ovarian endometrioma, as assessed with U/S performed prior to beginning r-hFSH treatment
* Severe endometriosis (American Fertility Society Classification Stage III or IV)
* World health organization (WHO) Group I anovulation
* Pelvic inflammatory disease within 1 year prior to beginning r-hFSH treatment
* Treatment with clomiphene citrate or gonadotrophins within 1 month prior to beginning r-hFSH treatment
* Abnormal undiagnosed gynecological bleeding
* Known allergy or hypersensitivity to human gonadotrophins preparations
* Known or current substance abuse
* Previous participation in this study or simultaneous participation in another clinical trial

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 1999-12; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | Day 4 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Ratio of ruptured follicles per follicle with diameter greater than or equal to (>=) 15 millimeter (mm) | Day 4 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Number of follicles with diameter greater than or equal to (>=) 11 millimeter (mm) | Day 4 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Ratio of ruptured follicles per follicle with diameter greater than or equal to (>=) 11 millimeter (mm) | Day 4 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])

SECONDARY OUTCOMES:
Percentage of participants with mono-follicular ovulation | Day 4 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Number of participants with biochemical pregnancy | Day 25-30 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Serum estradiol (E2) levels | Day 1, 2 and 6-9 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Serum androstenedione levels | Day 1, 2 and 6-9 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Serum total renin levels | Day 1, 2 and 6-9 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Serum vascular endothelial growth factor (VEGF) levels | Day 1, 2 and 6-9 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Endometrial thickness | Day 0, 1, 2, 3, 4 and 6-9 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Number of participants with clinical pregnancy | Day 25-30 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])
Serum progesterone (P4) levels | Day 1, 2 and 6-9 post r-hLH/u-hCG day (end of stimulation cycle [approximately 28 days])

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono International SA
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada